CLINICAL TRIAL: NCT06967207
Title: Electrical Impedance Tomography-Based Prognostic Model for ARDS: A Multicenter, Prospective, Observational Study
Brief Title: Electrical Impedance Tomography-Based Prognostic Model for ARDS
Status: Recruiting | Type: Observational
Sponsor: XiaoJing Zou,MD (Other)
Responsible Party: Sponsor-Investigator, XiaoJing Zou,MD, MD, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Other Study IDs: EIT20250331
Record Dates: First submitted 2025-04-22; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS); Ventilator-induced Lung Injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral whole blood samples will be collected and processed to isolate plasma, serum, and peripheral blood mononuclear cells (PBMCs). Processed samples (plasma, serum, PBMCs) will be stored at -80°C for future research. No DNA will be intentionally extracted or retained.

GROUPS / COHORTS (2):
- ARDS Patients for Training cohort: Training cohort
  Interventions: Other: Not applicable- observational study
- ARDS Patients for Validation cohort: Validation cohort
  Interventions: Other: Not applicable- observational study

INTERVENTIONS:
Other: Not applicable- observational study — Not applicable- observational study

SUMMARY:
This multicenter, prospective, observational study aims to develop and validate an EIT-based prognostic model for ARDS. By focusing on the pathophysiological characteristics of ARDS and the causes of ventilator-induced lung injury, the investigators intend to establish a prognostic model that reveals lung injury and heterogeneity, enabling risk stratification and guiding individualized treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the new 2023 ARDS global definition;
2. Age 18-80 years

Exclusion Criteria:

1. Expected death within 24 hours of screening;
2. Metastatic cancer (active malignancy with distant metastases);
3. Severe psychiatric disorders;
4. Pregnancy or postpartum status;
5. Pneumothorax or moderate to large pleural effusion without adequate drainage;
6. Chronic respiratory failure;
7. Patients with pulmonary embolism or pulmonary hypertension;
8. Heart failure patients: EF <50% or NYHA class III or IV;
9. Patient/family refusal to participate;
10. Participation in another interventional trial within 3 months prior to enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective, multicenter, observational cohort study that will enroll adult patients (aged 18-80 years) diagnosed with acute respiratory distress syndrome (ARDS) per the new 2023 ARDS global definition.
Sampling Method: Non-Probability Sample
Enrollment: 625 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
28-day mortality rate | From date of study enrollment (Day 0) until Day 28

SECONDARY OUTCOMES:
ICU mortality rate | From ICU admission to discharge, up to 24 weeks
60-day all-cause mortality rate | 60 days post-enrollment
90-day all-cause mortality rate | 90 days post-enrollment
Duration of mechanical ventilation (days) | From intubation to successful extubation, up to 28 days
Ventilator-free days (VFDs) at 28 days | 28 days post-enrollment
ICU length of stay (days) | From ICU admission to discharge, up to 24 weeks
Hospital length of stay | From hospital admission to discharge, up to 24 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Department of Critical Care Medicine, Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Department of Critical Care Medicine, Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Department of Critical Care Medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, China Department of, Wuhan, Hubei
  - Department of Emergency, Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes